CLINICAL TRIAL: NCT03194451
Title: Dental Stem Cells and Bone Tissue Engineering
Brief Title: Dental Stem Cells and Bone Tissue Engineering (CELSORDINO)
Acronym: CELSORDINO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-A00860-53/EUDRACT
Record Dates: First submitted 2017-06-16; First posted 2017-06-21 (Actual); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Tooth, Impacted
Keywords: bone tissue engineering, dental stem cell differentiation
MeSH Terms: conditions — Tooth, Impacted

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — teeth
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: non-interventional study — teeth collection

SUMMARY:
The main limitation in bone regeneration is the lack of vascularization of the newly shaped tissue. The main objective of this project is to check if the simultaneous differentiation of dental mesenchymal stem cells toward osteoblastic and endothelial lineage permits to obtain a new pre-vascularized tissue engineered bone construct.

We will then evaluate the boosting effect of the conditionned medium on cell differentiation and production of a prevascularized bone construct.

DETAILED DESCRIPTION:
This project aims to develop a new pre-vascularized tissue engineered bone construct, using human cells of a simple and non invasive tissue source: dental pulp.

We will isolate mesenchymal stem cells from dental tissue of wisdom teeth, extracted from patients aged between 13 and 17 years old.

The objectives are: (i) to assess in combination the endothelial differentiation and osteoblastic differentiation of dental pulp stem cells (immature third molar); (ii) to study the boosting effect of the conditionned medium on cell differentiation and production of a prevascularized bone construct.

The differentiation will be monitored by evaluation of biosynthesized matrix, bone mineralization (immunohistochimie, Westen Blot), histological response (Von Kossa, Alizarin Red) and presence and quantification of pseudo-vascular structures (angiogenesis assay), compared to reference value (commercial differentiation medium).

ELIGIBILITY:
Inclusion Criteria:

* patients aged between 13 and 17 years, who will come to Dental Service of University Regional Hospital Center of Nancy in order to have a tooth avulsion.
* patient who has received a complete information about research organization and who is not opposed to the use of his own data.
* patient who the representatives of parental authority have received a complete information about research organization and who are not opposed to the use of children's data.

Exclusion Criteria:

* patients with local or general pathology

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients aged between 13 and 17 years, who will be operated for wisdom tooth avulsion
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-07-10 (Estimated); Primary Completion 2017-08-20 (Estimated); Study Completion 2019-07-10 (Estimated)

PRIMARY OUTCOMES:
Bone mineralization | Day 28 of cell culture
  Measured parameter is equal or superior to reference value (commercial differentiation medium)

SECONDARY OUTCOMES:
presence and quantification of pseudo-vascular structures | Day 28 of cell culture
  Measured parameter is equal or superior to reference value (commercial differentiation medium)

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa MOBY, DD, PhD, Principal Investigator — IMoPA, UMR-CNRS 7365 CNRS-UL, Medicine Faculty

IPD SHARING:
Plan to Share IPD: No